CLINICAL TRIAL: NCT05803694
Title: ABL90 FLEX PLUS Clinical Precision Study for ctBil and FHbF Parameters in Neonatal Whole Blood
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-084471; 22003 (Other: Radiometer)
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2022-12

CONDITIONS: Blood Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples are collected to measure the ctBil and FHbF parameters in neonatal whole blood. Samples are destroyed when measurements are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ABL90 FLEX PLUS analyser running SW3.5 MR2. — The ABL90 FLEX PLUS analyzer is a portable, automated analyzer that measures pH, blood gases, electrolytes, metabolites, and oximetry in whole blood - utilizing 3 measuring modes (syringe, short probe, and capillary mode) to measure samples from a syringe, test tube or a capillary tube. The analyzer provides results for 17 parameters in 35 seconds using 65 μL heparinized whole blood.

SUMMARY:
Conducting the ABL90 FLEX PLUS Clinical Precision Study for ctBil and FHbF Parameters in Neonatal Whole Blood is to validate performance claims for precision of the ABL90 FLEX PLUS ctBil and FHbF parameters in neonatal whole blood while being influenced by testing environment that is representative of intended use environment, site variability, intended use testing environment and operator variability in a Point-of-Care (POC) setting.

The investigational device is the ABL90 FLEX PLUS incl. consumables, running SW3.5 MR2, manufactured by Radiometer Medical ApS.

The study is being conducted in Denmark and in total, a minimum of 54 subjects are to be enrolled to provide successful measurement values from 3 different sites.

DETAILED DESCRIPTION:
The conduct of the clinical study is to determine the repeatability of ctBil and FHbF parameters in neonatal whole blood using contrived fetal cord blood from umbilical cord/placenta measured by the intended users in syringe, short probe, and capillary modes available for ABL90 FLEX PLUS, in a POC setting.

The primary endpoint is the Repeatability (SD) for each parameter, parameter level and measuring mode, pooled across sites.

Participating sites are maternity wards or similar site conducting planned cesarean sections. Pregnant women 18 years of age or older admitted to the maternity ward to undergo cesarian section after week 38 of gestation will be enrolled in the clinical study. When the subject has signed ICF, the site will collect cord blood from umbilical cord/placenta and when relevant prepare contrived samples by having access to adult type 0 Rh neg whole blood for diluting HbF in cord blood.

Three POC users, such as a nurse, a physician, or a therapist that care for the woman in the maternity ward will perform all measurements and they shall contribute evenly to the total number of samples measured. Replicate measurements shall be performed by the same user.

6-10 mL of cord blood is collected in a blood collection syringe from each umbilical cord/placenta, contrived, and the sample is aliquoted into 5 safePICO aspirators (max volume 1.5 mL) or into 25 capillary tubes.

At each site, samples will be collected for the 2 parameters, 3 modes and 3 levels, completing measurements from minimum of 18 samples from 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age or older admitted to the maternity ward to undergo cesarian section.
* Informed consent collected from subject able to understand information given, and willing and able to voluntarily give their consent to participate in this study.
* Subject evaluated by the principal investigator or designee as suitable for the study according to the protocol.

Exclusion Criteria:

* Subjects with known infectious disease such as Hepatitis C or HIV (to ensure the operator safety).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant women 18 years of age or older admitted to the maternity ward to undergo cesarian section after week 38 of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
ABL90 FLEX PLUS Clinical Precision | 5 hours
  Repeatability (SD) for each parameter (ctBil and FHbF), parameter level and measuring mode, pooled across sites.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Radiometer Medical, Copenhagen, Brønshøj
  - Ellen Løkkegaard, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
When the Clinical Study Report has been finalized, Data result will be available for public on platforms and in articles.
Supporting Information: CSR
Time Frame: January 2025